CLINICAL TRIAL: NCT05126719
Title: An Open-Label, Multi-Center Phase II Clinical Study to Evaluate the Efficacy and Safety of MRG003 in Patients With Recurrent Metastatic Nasopharyngeal Carcinoma
Brief Title: A Study to Evaluate the Efficacy and Safety of MRG003 in Patients With Recurrent Metastatic Nasopharyngeal Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Miracogen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MRG003-005
Record Dates: First submitted 2021-11-17; First posted 2021-11-19 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Recurrent or Metastatic Nasopharyngeal Carcinoma
Keywords: MRG003; Antibody Drug Conjugate (ADC); Nasopharyngeal Carcinoma.; EGFR
MeSH Terms: conditions — Recurrence; Nasopharyngeal Carcinoma | interventions — Capecitabine; Docetaxel

STUDY DESIGN:
Intervention Model Description: The study consists of two stages. Part A of this study is a single arm IIa clinical study and Part B is a parallel IIb study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MRG003 (Experimental): Part A: On the first day of every 3 weeks, MRG003 will be administered via intravenous infusion at 2.0 mg/kg or 2.3 mg/kg calculated based on the actual body weight.
  Part B: On the first day of every 3 weeks, MRG003 will be administered via intravenous infusion at 2.3 mg/kg calculated based on the actual body weight.
  Interventions: Drug: MRG003
- Capecitabine tablets/Docetaxel injection (Active Comparator): Part B: Capecitabine tablets: 1000 mg/m2, bid, d1-14, po, Q3W, or Docetaxel injection: 75 mg/m2, d1, IV, Q3W
  Interventions: Drug: Capecitabine tablets; Drug: Docetaxel injection

INTERVENTIONS:
Drug: MRG003 — Administered intravenously
  Arms: MRG003
Drug: Capecitabine tablets — Administered peros
  Arms: Capecitabine tablets/Docetaxel injection
Drug: Docetaxel injection — Administered intravenously
  Arms: Capecitabine tablets/Docetaxel injection

SUMMARY:
The objective of this study is to assess the safety, efficacy, pharmacokinetics, and immunogenicity of MRG003 in patients with recurrent metastatic nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
The study consists of two stages.

Part A of this study is an open-label, single arm, multicenter Phase IIa clinical study in patients with inoperable, radiotherapy ineligible RM-NPC who have failed (or are intolerable) at least 1 prior line platinum-based systemic chemotherapy and PD-1 (L1) inhibitors.

Part B is an open-label, randomized, multicenter Phase IIb study to compare the efficacy and safety of MRG003 versus capecitabine/docetaxel in patients with RM-NPC who have failed at least 2 prior lines of systemic chemotherapy and PD-1 (L1) inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Willing to sign the ICF and follow the requirements specified in the protocol.
* Age: ≥18 years, ≤75 years
* Expected survival time>3 months.
* Patients with histologically confirmed unresectable, radiation-ineligible recurrent metastatic nasopharyngeal carcinoma.
* Part A: Metastatic nasopharyngeal carcinoma that has failed or recurred or was intolerant to at least 1 prior line platinum-based systemic chemotherapy and PD-1/PD-L1 inhibitors
* Part B: have documented failure of at least 2 prior lines of PD-1 (L1) and therapysystemic chemotherapy, which include at least platinum-based regimen, gemcitabine, taxanes/capecitabine.
* Patients must have measurable lesions according to the Response Evaluation Criteria in Solid Tumors (RECIST v1.1).
* ECOG performance score 0 or 1.
* Organ functions and coagulation function must meet the basic requirements.
* No severe cardiac dysfunction with left ventricular ejection fraction (LVEF) ≥ 50%.
* Serum or urine pregnancy test negative within 72 hours before the first dose of investigational drug.
* Patients with childbearing potential must use effective contraception during the treatment and for 6 months after the last dose of treatment.

Exclusion Criteria:

* Grade ≥2 peripheral neuropathy per CTCAE v5.0.
* Is expected to require surgery or any other form of systemic or local anti-tumor therapy during the study.
* Received systemic chemotherapy, targeted therapy, biologics or immunotherapy, or major surgery (except for minor surgery within 2 weeks and fully recovered) within 3 weeks prior to the first dose of study treatment; received thoracic radiotherapy >30 Gy within 6 months prior to the first dose of study treatment; received prior radiotherapy (except radiotherapy for CNS, wash-out period ≥ 28 days is required) within 14 days before the first dose of study treatment, received traditional Chinese medicine with anti-tumor indications within the 2 weeks before the first dose of study treatment.
* Known active central nervous system (CNS) metastases and/or meningeal metastases. Patients with brain metastases may participate provided they are treated and stable
* Residual toxicities due to prior anti-tumor therapy (including biologics, targeted therapy, immunotherapy, chemotherapy or radiotherapy) or ≥ Grade 1 (CTCAE v5.0) clinically significant laboratory abnormality.
* History of severe cardiac dysfunction, stroke, or transient ischemic attack (TIA) within 6 months prior to enrollment. History of ventricular tachycardia or torsades de pointes. Any clinically important abnormality in the rhythm, conduction, or morphology of the resting ECG. Note: Patients with arrhythmia are eligible if they are receiving antiarrhythmic medication and the screening electrocardiogram (ECG) shows controllable rhythm and heart rate.
* Pulmonary embolism or deep venous thrombosis within 3 months prior to the first dose of study drug.
* Known history of malignancy (except for patients with cutaneous basal cell carcinoma, superficial bladder carcinoma, cutaneous squamous cell carcinoma, cervical carcinoma in situ, or papillary thyroid carcinoma who have undergone successful curative treatment) unless the patient has received potentially curative therapy and has not had disease recurrence within 5 years starting from the treatment.
* Note: The 5-year recurrence-free time requirement does not apply to NPC for which the patient is enrolled.
* Uncontrolled or poorly controlled hypertension (e.g., systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg) or diabetes mellitus (glycosylated hemoglobin (HbA1c) > 8%).
* Patients with active bleeding, history of coagulopathy, or receiving coumarin anticoagulant therapy.
* History of ≥ Grade 3 immune-related AEs (irAEs), including skin toxicity, diarrhea, enteritis, fatigue, immune-related nephritis, immune-related hepatitis, and infusion reactions.
* Known allergic reactions to any component or excipients of MRG003 (citric acid monohydrate, sodium citrate dihydrate, trehalose dihydrate, sodium chloride, and polysorbate 80) or capecitabine/docetaxel, or known allergic reactions to other anti-EGFR agents (including investigational drug) or to other monoclonal antibodies ≥ Grade 3.
* Known active hepatitis B or C. Presence of other serious liver diseases, including chronic autoimmune hepatic disorders, primary biliary cirrhosis or sclerosing cholangitis, alcoholic liver disease, or nonalcoholic steatohepatitis (NASH).
* Concurrent, serious, uncontrolled infection or known infection with human immunodeficiency virus (HIV) (HIV antibody positive), or diagnosis of acquired immunodeficiency syndrome (AIDS); or uncontrolled autoimmune disease; or previous allogeneic tissue/organ transplantation, stem cell or bone marrow transplantation, or previous solid organ transplantation.
* Active bacterial, viral, fungal, rickettsial, or parasitic infection requiring systemic anti-infection therapy (unless treated and resolved prior to study treatment).
* Received live-virus vaccines within 30 days prior to the first dose of study treatment. Seasonal influenza vaccines or approved COVID-19 vaccines that do not contain live virus are permitted.
* History of moderate to severe dyspnea at rest or severe primary lung disease (current need for continuous oxygen therapy and oxygen saturation < 93% without oxygen therapy) due to advanced cancer or its complications, or history of any interstitial lung disease (ILD) (including ILD that requires oral or intravenous corticosteroids) or noninfectious pneumonitis
* Patients who are receiving an immunologically based treatment for any reason, including chronic use of systemic steroids equivalent to > 10 mg/day of prednisone within 7 days prior to the first dose of study treatment or at any time during the study. Note: Use of inhaled or topical steroids or systemic corticosteroids equivalent to ≤ 10 mg/day prednisone is permitted, as is short-term use of corticosteroids at doses equivalent to > 10 mg/day prednisone (e.g., pre-medication prior to contrast).
* Chronic autoimmune or inflammatory disease requiring or receiving systemic therapy within the last 2 years, including but not limited to inflammatory bowel disease, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, Wegener's granulomatosis, Sjogren's syndrome, Guillain - Barre's syndrome, multiple sclerosis, vasculitis, or glomerulonephritis (exceptions: vitiligo, hypothyroidism on stable hormone replacement therapy, controlled asthma, type I diabetes mellitus, Graves' disease, Hashimoto's disease, or with medical monitor's approval).
* Uncontrolled pleural, abdominal, pelvic effusion or pericardial effusion that requires ≥ 1 drainage per month.
* Patients who are using strong CYP3A4 inhibitors or inducers and for who stop the use is not recommended.
* Any patient with a positive pregnancy or is breast-feeding. Female and male patients who are not expected to use adequate contraception during treatment and for 180 days after the last dose of treatment.
* Any other disease or clinically significant abnormality in laboratory parameters, or serious medical or psychiatric illnesses/conditions, substance abuse disorder including alcoholism, which in the judgment of the Investigator might compromise the safety of the patient, integrity of the study, interfere with the patient participation in the study, or confound or compromise the study objectives and their interpretability.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2023-04-06 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) by Independent Review Committee (IRC) | Baseline to disease progression, intolerable drug-related toxicities, withdrawal of consent, or study discontinuation for any reasons (up to 24 months)
  ORR is defined as the proportions of patients with a complete response (CR) and partial response (PR). ORR will be assessed by Independent Review Committee (IRC) according to RECIST v1.1.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) by Investigator | Baseline to Baseline to disease progression, intolerable drug-related toxicities, withdrawal of consent, or study discontinuation for any reasons (up to 24 months)
  ORR is defined as the proportions of patients with a complete response (CR) and partial response (PR). ORR will be assessed by investigator according to RECIST v1.1.
Progression Free Survival (PFS) | Baseline to Baseline to disease progression, intolerable drug-related toxicities, withdrawal of consent, or study discontinuation for any reasons (up to 24 months)
  PFS is defined as the duration from the start of treatment or randomization (part B) to the onset of tumor progression or death of any cause.
Duration of Response (DoR) | Baseline to Baseline to disease progression, intolerable drug-related toxicities, withdrawal of consent, or study discontinuation for any reasons (up to 24 months)
  DOR is defined as the duration from the initial recording of objective disease response to the first onset of tumor progression, or death of any cause.
Disease Control Rate (DCR) | Baseline to Baseline to disease progression, intolerable drug-related toxicities, withdrawal of consent, or study discontinuation for any reasons (up to 24 months)
  DCR is defined as the proportions of patients achieving CR, PR, and stable disease (SD) after treatment.
Overall Survival (OS) | Sign the informed consent form to Baseline to disease progression, intolerable drug-related toxicities, withdrawal of consent, or study discontinuation for any reasons (up to 24 months)
  OS is defined as the duration from the start of treatment or randomization (part B) to death of any cause.
Adverse Events (AEs) | Baseline to 30 (for AE) and 45 (for SAE) days after the last dose of study treatment.
  Any reaction, side effect, or untoward event that occurs during the course of the clinical trial whether or not the event is considered related to the study drug.
PK parameter for MRG003: (Cmax) | Baseline to 30 days after the last dose of study treatment
  Maximum observed plasma concentration.
PK parameter for MRG003: (AUClast) | Baseline to 30 days after the last dose of study treatment.
  Area under the curve up to the last validated measurable plasma concentration.
PK parameter for total antibody (TAb): Cmax | Baseline to 30 days after the last dose of study treatment.
  Maximum observed plasma concentration.
PK parameter for TAb: AUClast | Baseline to 30 days after the last dose of study treatment.
  Area under the curve up to the last validated measurable plasma concentration.
PK parameter for Monomethyl Auristatin E (MMAE): Cmax | Baseline to 30 days after the last dose of study treatment.
  Maximum observed plasma concentration.
PK parameter for MMAE: AUClast | Baseline to 30 days after the last dose of study treatment.
  Area under the curve up to the last validated measurable plasma concentration.
The proportion of patients with positive ADA immunogenicity results. | Baseline to 30 days after the last dose of study treatment.
  The incidence of patients with positive ADA immunogenicity results per each pre-specified time point.

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, Doctor, Principal Investigator — Sun Yat-sen University
Locations (23):
- China (23):
  - Peking University Cancer Hospital, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Maoming People's Hospital, Maoming, Guangdong
  - Cancer Hospital of Shantou University Medical College, Shantou, Guangdong
  - Yue Bei People's Hospital, Shaoguan, Guangdong
  - Zhongshan City People's Hospital, Zhongshan, Guangdong
  - Guigang City People's Hospital, Guigang, Guangxi
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning, Guangxi
  - People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - The Affiliated Cancer Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Hainan General Hospital, Haikou, Hainan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - First Affiliated Hospital of Gannan Medical University, Ganzhou, Jiangxi
  - Ganzhou Cancer Hospital, Ganzhou, Jiangxi
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - Yibin Second People's Hospital, Yibin, Sichuan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No